CLINICAL TRIAL: NCT01182142
Title: Phase II Study of Capecitabine in Metastatic Non-clear Cell Renal Cell Carcinoma Patients
Brief Title: Study of Capecitabine in Metastatic Non-clear Cell Renal Cell Carcinoma (RCC) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Lev Demidov, N.N. Blokhin Russian Cancer Research Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRT-06.CAP
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine (Experimental): All patients will receive capecitabine.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — 1,250 mg/m2 orally twice a day, days 1-14

SUMMARY:
Capecitabine is an orally-administered chemotherapeutic agent used in the treatment of metastatic breast and colorectal cancers. The role of capecitabine in treatment of metastatic renal cell carcinoma is discussed. In this trial, we are evaluating efficacy of capecitabine in metastatic renal cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed non-clear cell renal cell carcinoma
* confirmed metastatic sites
* no chemotherapy in history

Exclusion Criteria:

* metastases in CNS
* previous targeted therapy
* other tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 12 months

SECONDARY OUTCOMES:
Overall survival Progression-free survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lev Demidov, MD, D.Sc., Principal Investigator — N.N. Blokhin Russian Cancer Research Center
Locations (1):
- Natalia Petenko, Moscow, Russia

REFERENCES:
- [Derived] Tsimafeyeu I, Demidov L, Kharkevich G, Petenko N, Galchenko V, Sinelnikov I, Naidzionak U. Phase II, multicenter, uncontrolled trial of single-agent capecitabine in patients with non-clear cell metastatic renal cell carcinoma. Am J Clin Oncol. 2012 Jun;35(3):251-4. doi: 10.1097/COC.0b013e31820dbc17. PMID 21358295
- See also: Related Info — http://www.ronc.ru/